CLINICAL TRIAL: NCT05262413
Title: A Study of QL1706 Plus Lenvatinib in Subjects With Advanced Renal Cell Carcinoma(RCC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-107
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Advanced Renal Cell Carcinoma
Keywords: QL1706
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QL1706 Plus Lenvatinib (Experimental): QL1706 5mg/kg administered intravenously (IV), every 3 weeks, plus Lenvatinib 20 mg or 14mg administered orally, once daily.
  Interventions: Drug: QL1706 Plus Lenvatinib

INTERVENTIONS:
Drug: QL1706 Plus Lenvatinib — QL1706 5mg/kg administered intravenously (IV), every 3 weeks, plus Lenvatinib 20 mg or 14mg administered orally, once daily.
  Other Names: PSB205

SUMMARY:
This is a phase 1b, multicenter, open label, single arm study designed to evaluate the efficacy, safety, tolerability, pharmacokinetic (PK), and immunogenicity of QL1706 plus lenvatinib in subjects with advanced RCC.

DETAILED DESCRIPTION:
This study included a screening period, a treatment period, and a post-treatment follow-up period. Safety will be monitored throughout the study. At the same time, the pharmacokinetics and immunogenicity of QL1706 and lenvatinib in subjects with advanced renal cell carcinoma were evaluated, and the preliminary efficacy of QL1706 combined with lenvatinib in subjects with advanced renal cell carcinoma was evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects participate voluntarily and sign informed consent.
2. Male or female subjects aged 18 years or older.
3. Pathological confirmation of renal cell carcinoma (RCC) mainly with a clear-cell component
4. At least 1 measurable target lesion according to Response Evaluation in Solid Tumors (RECIST) 1.1
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. Life expectancy of ≥6 months.
7. The functional level of important organs must meet the requirements before the first dose of study drug.
8. Male and female patients able to have children must agree to use highly effective method of contraception throughout the study and for at least 180 days after last dose. Female subjects who are not pregnant or breastfeeding.
9. Before the first use of the investigational drug, all the reversible toxicity of the previous antitumor therapy returned to ≤1 (according to CTCAE V5.0),Excluding any grade of hair loss and pigmentation, grade 2 or less peripheral sensory neuropathy, and other abnormalities that the investigator and/or sponsor assessed to outweigh the risk of toxicity.

Exclusion Criteria:

1. Symptomatic central nervous system (CNS) metastasis, leptomeningeal metastasis or spinal cord compression due to metastasis before the first dose of study drug.
2. Received radiotherapy or other local treatment within 2 weeks before the first dose of study drug, and did not recover from the adverse reactions of local treatment.
3. Patients with a history of other malignant tumors within 5 years before signing the informed consent.
4. Active autoimmune diseases that exist within 2 years prior to the first dose of study drug and require systemic treatment.
5. Hypertension uncontrolled by 2 or more antihypertensive drugs (BP ≥150/90 mmHg at Screening).
6. Previous history of hypertensive crisis or hypertensive encephalopathy.
7. History of allogeneic hematopoietic stem cell transplantation or organ transplantation (except corneal transplantation)
8. Were receiving long-term systemic steroid therapy within 7 days prior to first dose of the study drug.
9. HIV-positive patients; known to have received anti-tuberculosis therapy within one year before the first study treatment; hepatitis B surface antigen (HBsAg) positive and hepatitis B virus deoxyribonucleic acid (HBV DNA) ≥ 2000 IU/ml or 104 copies/ml ; HCV antibody positive and HCV RNA positive.
10. HbsAg and anti-HCV antibodies were positive.
11. Patients with active pulmonary tuberculosis within one year before the first use of the investigational drug.
12. Subjects with any of the cardiovascular diseases were excluded as defined.
13. The patient is known to have a history of psychotropic substance abuse, alcoholism, or drug use; a clear history of neurological or psychiatric disorders, including epilepsy or dementia or hepatic encephalopathy.
14. Participants who participated in other clinical studies and used other study drugs within 4 weeks before the first dose of study drug.
15. Known history of hypersensitivity to macromolecular protein preparation or any components of the the study drugs.
16. Received a live vaccine within 4 weeks prior to the first dose of study drug.
17. Major surgery within 4 weeks prior to first use of the study drug.
18. Past and/or current history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, severely impaired lung function, etc. may interfere with the detection and management of suspected drug-related pulmonary toxicity.
19. Arteriovenous thromboembolic events, including cerebrovascular accident or history of stroke or transient ischemic attack, pulmonary embolism, deep vein embolism, or other serious thromboembolic events within 6 months prior to the first use of the investigational drug.
20. Patients at risk of severe perforation or bleeding.
21. Clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of the study drug.
22. Gastrointestinal perforation, gastrointestinal or non-gastrointestinal fistula, or abdominal abscess within 6 months prior to first dose of the study drug.
23. Any life-threatening bleeding event within 3 months prior to the first trial drug, including the need for blood transfusion therapy, surgery or topical therapy, ongoing drug therapy.
24. Concomitant treatment with therapeutic doses of anticoagulants, such as heparin, thrombin, or factor Xa inhibitors, or antiplatelet drugs.
25. Patients who, in the investigator's judgment, may increase the risks associated with the study, may interfere with the interpretation of the study results, or are deemed unsuitable for enrollment by the investigator and/or sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-28 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Up to approximately 2 years
  Safety and tolerability, as defined by the rate of treatment-related adverse events as assessed by NCI CTCAE v5.0